CLINICAL TRIAL: NCT05089071
Title: Effect of Two Colonoscopy AI Systems for Colon Polyp Detection According to the False Positive Rates of the Systems: A Single-center Prospective Study
Brief Title: Effect of Two Colonoscopy AI Systems for Colon Polyp Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SNUH IRB 2107-235-1240
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-03

CONDITIONS: Adenoma; Colonoscopy; Sessile Serrated Adenoma
Keywords: endoscopist; adenoma detection rate; colonoscopy; artificial intelligence
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Intervention Model Description: The primary outcome was the comparison of ADR between the control and AI groups according to the intervention system (SCAI vs ENAD system).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CADe group (Experimental): Endoscopists perform colonoscopy with CADe system
  Interventions: Device: Assist by artificial intelligence system for colon polyp detection
- Control (No Intervention): Endoscopists perform colonoscopy without CADe system

INTERVENTIONS:
Device: Assist by artificial intelligence system for colon polyp detection — Assist by artificial intelligence system for colon polyp detection
  Arms: CADe group

SUMMARY:
Computer-aided detection (CADe) systems have been actively researched for polyp detection in colonoscopy. The investigators aim to identify the effect of two CADe systems according to the system performance on false positive rate

DETAILED DESCRIPTION:
Artificial intelligence technology based on deep learning is being applied in various medical fields, and research is being actively conducted to develop computer-aided detection (CADe) systems for colonoscopies to overcome the limitation of the variance of human skills. These well-trained CADe systems demonstrated high performance for neoplastic polyp detection and reported a 44% increase in adenoma detection rate (ADR) for endoscopists. However, the level of performance in the CADe system is not clear for expert endoscopists to be useful for ADR increase.

Furthermore, false positives(FPs) of the CADe system may negatively influence ADR during a screening colonoscopy. Accordingly, the investigators sought to identify the effect of the colonoscopy CADe system according to FP performance in endoscopists with various levels. The investigators hypothesized that the CADe system with low FPs would be useful to prevent the decrease in ADR in case of a high endoscopy workload according to the performance of CADe systems.

ELIGIBILITY:
Inclusion Criteria:

patient for screening or surveillance colonoscopy patients agreed with participating in the study

Exclusion Criteria:

patients who do not agree with participating in the study patients with a history of colon resection patients with a history of inflammatory bowel resection patients with poor bowel preparation

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3046 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 12 months
  proportion of colonoscopies with at least one adenoma detected overall and as detected by the physician.
Sessile serrated lesion detection rate | 12 months
  proportion of colonoscopies with at least one sessile serrated lesion detected overall and as detected by the physician.

SECONDARY OUTCOMES:
polyp detection rate | 12 months
  proportion of colonoscopies with at least one polyp detected overall and as detected by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Ho Bae, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Healthcare System Gangnam Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963